CLINICAL TRIAL: NCT01825603
Title: A Phase I Study of ADH-1 and Gemcitabine Plus Cisplatin in Patients With Unresectable or Metastatic Pancreatic and Biliary Tract Cancers
Brief Title: ADH-1, Gemcitabine Hydrochloride & Cisplatin in Treating Metastatic Pancreatic or Biliary Tract Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Adherex Technologies, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0470-12-FB; NCI-2013-00406 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA036727 (NIH); P50CA127297 (NIH)
Record Dates: First submitted 2013-03-27; First posted 2013-04-05 (Estimated); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Ampulla of Vater Adenocarcinoma; Gallbladder Adenocarcinoma; Metastatic Pancreatic Adenocarcinoma; Pancreatic Adenocarcinoma; Stage III Ampulla of Vater Cancer; Stage III Intrahepatic Cholangiocarcinoma; Stage III Pancreatic Cancer; Stage IIIA Gallbladder Cancer; Stage IIIA Hilar Cholangiocarcinoma; Stage IIIB Gallbladder Cancer; Stage IIIB Hilar Cholangiocarcinoma; Stage IV Ampulla of Vater Cancer; Stage IVA Gallbladder Cancer; Stage IVA Hilar Cholangiocarcinoma; Stage IVA Intrahepatic Cholangiocarcinoma; Stage IVA Pancreatic Cancer; Stage IVB Gallbladder Cancer; Stage IVB Hilar Cholangiocarcinoma; Stage IVB Intrahepatic Cholangiocarcinoma; Stage IVB Pancreatic Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Pancreatic Neoplasms; Gallbladder Neoplasms; Klatskin Tumor | interventions — N-Ac-CHAVC-NH2; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ADH-1, cisplatin, gemcitabine hydrochloride) (Experimental): Patients receive ADH-1 IV over 20-80 minutes on days 1, 4, 8, 11, 15, and 18, cisplatin IV and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responsive disease may receive maintenance therapy with cisplatin and gemcitabine hydrochloride.
  Interventions: Drug: ADH-1; Drug: Cisplatin; Drug: Gemcitabine Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: ADH-1 — Given IV
  Other Names: Exherin
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of ADH-1 when given together with gemcitabine hydrochloride and cisplatin in treating patients with pancreatic or biliary tract cancer that has spread from where it started to nearby tissue or lymph nodes (locally advanced) or spread to other parts of the body (metastatic) and cannot be removed by surgery. ADH-1 may stop the growth of cancer cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as gemcitabine hydrochloride and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ADH-1 together with gemcitabine hydrochloride and cisplatin may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the toxicities and determine the recommended dose of ADH-1 given twice weekly for 3 weeks in combination with cisplatin and fixed-dose rate gemcitabine (gemcitabine hydrochloride) given on weeks 1 and 2 of the 3 week schedule for 3 cycles in patients with locally advanced or metastatic pancreatic or biliary tract adenocarcinomas.

SECONDARY OBJECTIVES:

I. To evaluate changes in the levels of intercellular adhesion molecule 1 (ICAM-1), E-selectin, vascular endothelial growth factor (VEGF), soluble vascular endothelial growth factor receptor (VEGFR) and basic fibroblast growth factor (B-FGF) during therapy with ADH-1, cisplatin and gemcitabine.

II. Radiographic assessment of disease status after 3 cycles of chemotherapy with ADH-1, cisplatin and gemcitabine.

III. To evaluate progression-free and overall survival of patients with locally advanced or metastatic pancreatic or biliary tract adenocarcinomas treated with ADH-1 given with cisplatin and fixed dose rate gemcitabine for 3 cycles. Patients with stable or responsive disease after 3 cycles will continue on maintenance cisplatin and fixed dose rate gemcitabine.

OUTLINE: This is a dose-escalation study of ADH-1.

Patients receive ADH-1 intravenously (IV) over 20-80 minutes on days 1, 4, 8, 11, 15, and 18, cisplatin IV and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responsive disease may receive maintenance therapy with cisplatin and gemcitabine hydrochloride.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have adenocarcinoma of the pancreas or biliary tree (intrahepatic or extrahepatic cholangiocarcinoma, gallbladder or ampulla of Vater) that is locally advanced, but non-resectable, metastatic or residual disease after attempted surgical resection
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 or better
* Absolute neutrophil count (ANC) of 2000 per mcL or higher
* Platelet count of 100,000 per mcL or higher
* Patients must have a serum creatinine that is at or below the upper limits of the institutional normal range OR a creatinine clearance of 60 mL per min or higher corrected for body surface area (BSA)
* The total bilirubin must be at or below 2.0 mg/dL in the absence of biliary obstruction; if the patient has biliary obstruction, biliary decompression will be required; either endoscopic placement of a biliary stent or percutaneous transhepatic drainage is acceptable; once biliary drainage has been established, institution of protocol therapy may proceed when the total bilirubin falls to 3.0 mg/dL or lower
* Patients need not have measurable disease for this study
* The patient must be aware of the neoplastic nature of his/her disease and willingly provide written, informed consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts
* Women of reproductive potential must be non-pregnant and non-nursing and must agree to employ an effective barrier method of birth control throughout the study and for up to 6 months following treatment
* Women of child-bearing potential must have a negative pregnancy test within 7 days of initiating study; (no childbearing potential is defined as age 55 years or older and no menses for two years or any age with surgical removal of the uterus and/or both ovaries)

Exclusion Criteria:

* Patients may not have received prior chemotherapy for metastatic adenocarcinoma of the pancreas or biliary tract; prior adjuvant chemotherapy is acceptable provided that 6 months or longer has elapsed since completion of the prior therapy
* History of allergy to platinum compounds or to antiemetics appropriate for administration in conjunction with protocol-directed chemotherapy
* Uncontrolled inter-current illness including, but not limited to ongoing or active infection requiring intravenous antibiotics, symptomatic congestive heart failure, unstable angina pectoris, or serious, uncontrolled cardiac arrhythmia, that might jeopardize the ability of the patient to receive the chemotherapy program outlined in this protocol with reasonable safety
* Pregnant and nursing women are excluded from this study
* Patients with prior malignancy will be excluded except for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas, or other cancers from which the patient has been disease-free for at least 5 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Recommended dose of ADH-1, defined as the highest dose tested which results in dose-limiting toxicities in no more than 1 of 6 evaluable patients based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | 21 days
  The incidence rates of adverse events will be described by dose level. The frequency of occurrence of overall toxicity, categorized by toxicity grades, will be described.

SECONDARY OUTCOMES:
Changes in the levels of ICAM-1, E-selectin, VEGF, soluble VEGFR and B-FGF | After all patients complete cycle 1, about 2 years after initial patient enrolled
  Summarized using descriptive statistics
Progression-free survival | From the first date of therapy until the first notation of clinical progression, relapse or death from any cause, assessed up to 2 years
  Plotted following the method of Kaplan and Meier.
Survival | From the first date of therapy until the date of death from any cause, assessed up to 2 years
  Plotted following the method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Overall Officials: Jean L Grem, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States